CLINICAL TRIAL: NCT04765098
Title: A Randomized Controlled Trial of Tamoxifen Versus Etoposide for Patients With First Recurrence of Glioblastoma Multiforme
Brief Title: Tamoxifen Versus Etoposide After First Recurrence in GBM Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0014
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Tamoxifen; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoposide (Active Comparator)
  Interventions: Drug: Etoposide
- Tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen 20 mg daily for 3 days then 20 mg BID for 3 days then increase by 20 mg daily every 3 days until 100 mg BID continuously
  Arms: Tamoxifen
Drug: Etoposide — etoposide 50mg/m2 daily
  Arms: Etoposide

SUMMARY:
The investigator propose a single-center randomized phase II controlled study designed to compare the management of first recurrence of GBM using etoposide versus tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven GBM with progression after previous first line chemoradiotherapy with temozolomide.
2. Progression documented by MRI with at least one bi-dimensionally measurable target lesion with one diameter of at least 10 mm, visible on two or more axial slices 5 mm apart.
3. Not received radiotherapy within the three months before the diagnosis of progression.
4. Stable or decreasing dose of corticosteroids prior to randomization: corticosteroids (dexamethasone) should be given at the lowest dose needed to control symptoms arising from increased intracerebral edema.
5. ECOG performance 0-2 (Appendix 2).
6. Age from 18-65 years.
7. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
8. Patients of childbearing / reproductive potential should use adequate birth control methods, as defined by the investigator, during the study treatment period and for a period of 60 days after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
9. Laboratory evaluation obtained within 7 days prior to randomization, with adequate function as defined below:

   * ANC ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Serum creatinine ≤ 1.5 times ULN
   * Total serum bilirubin ≤ 1.5 times ULN
   * ALT < 3 times ULN
   * AST < 3 times ULN
   * Alkaline phosphatase < 3 times ULN
10. Patient must understand and sign an informed consent prior to study registration.

Exclusion Criteria:

1. History of another malignancy or a concurrent malignancy (exceptions include patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
2. Uncontrolled hypertension (systolic blood pressure >150 mm Hg or diastolic blood pressure >100 mm Hg).
3. Any arterial or venous thrombosis up to 6 months before registration.
4. Evidence of recent hemorrhage on brain MRI.
5. Substantial cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
3 month progression-free survival | 3 months
  Time between randomization and radiographic or clinical progression leading to change in therapy for recurrent disease or death due to any cause.

SECONDARY OUTCOMES:
One-year progression-free survival | 12 months
  Time between randomization and radiographic or clinical progression leading to change in therapy for recurrent disease or death due to any cause.
Overall survival | Median, 6-month, 1-year, and 2-year OS rates will be measured
  Time between randomization and death due to any cause. Patients without an event will be censored the last time they were known to be alive.
Health-related quality-of-life status | Throughout study completion, up to 5 years.
  Health-related quality-of-life will be assessed using the EORTC QLQ-BN20 brain tumor module questionnaire. This is a self-report questionnaire consisting of 20 items that assess future uncertainty, visual disorder, motor dysfunction, and communication deficit in brain tumor patients
Adverse events | Throughout the whole duration of the trial, up to 5 years
  This includes fatigue, hematologic toxicities (neutropenia, thrombocytopenia, leukopenia, anemia), liver toxicities, hypertension, diarrhea, seizures and thrombosis and will all be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada